CLINICAL TRIAL: NCT05917132
Title: Production of Gut Microbiota-Derived Metabolites in Response to Different Fatty Acid Profiles
Acronym: METAc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Alain Veilleux, Professor, Laval University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-109
Record Dates: First submitted 2023-06-15; First posted 2023-06-23 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Obesity, Abdominal; Diabete Type 2
Keywords: Gut Microbiome; Endocannabinoidome; Metabolites; Microbiome-Endocannabinoidome Axis; Obesity; Type 2 Diabetes; Nutrition; Fatty Acids
MeSH Terms: conditions — Obesity, Abdominal; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single (Experimental): All participating subjects will undergo 3 feeding phases : 3 days of a run-in diet, 2 days of a polyunsaturated fatty acid (PUFA) diet and 2 days of a saturated fatty acid (SFA) diet.
  Interventions: Other: Nutritionnal intervention

INTERVENTIONS:
Other: Nutritionnal intervention — Participants will be provided with meals corresponding to each diet during the week. Participants will be required to eat only the meals provided.

SUMMARY:
The proposed project mainly aims to investigate the microbial processes leading to dietary metabolites production, independently of long-term microbiota adaptation to the diet, by measuring the microbiota-derived metabolite production from a meal sequence rich in saturated fatty acids (SFA) or the same meals but rich in polyunsaturated fatty acids (PUFA) in individuals with or without obesity and Type 2 diabetes (T2D)

DETAILED DESCRIPTION:
The gut microbiota interacts with the host's enteric and systemic functions through the production of gut microbiota-derived metabolites. A subset of these metabolites, the endocannabinoids (eCB) and their congeners are derived from fatty acids and play a crucial role in metabolic health.

The research project aims to study gut microbiota-derived metabolites, including the eCB and their congeners, in response to a 2-day diet rich in polyunsaturated fatty acids or rich in saturated fatty acids in individuals with or without abdominal obesity and type 2 diabetes.

The investigators hope to better understand the kinetic production of circulating endocannabinoidome mediators derived from fatty acids in the diet.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 45 and 65 years, menopaused women ;
* Body mass index between 20 to 35 kg/m² ;
* General good health ;
* Score of diet quality (HEI) between 40 and 70 ;
* Computer and Internet access ;
* Basic understanding of written French ;
* Daily stool frequency.

Exclusion Criteria:

* Intestinal pathologies including inflammatory bowel disease and gastrointestinal cancers ;
* Alcohol consumption greater than 15 portions for men and 10 for women weekly.
* Active tobacco and cannabis usage ;
* Consumption of omega-3 dietary supplements ;
* Consumption of dietary supplements (vitamins and probiotics) - must be ceased 2 weeks before the dietary intervention ;
* Completion of a course of antibiotics in the past 3 months ;
* Important weight change (+/- 5 kg) in the past 6 months ;
* Type 1 diabetes or insulin-treated diabetes.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Fasting and postprandial lipid metabolite production in response to dietary lipid intervention in abdominal obesity and type 2 diabetes | 7 days
  Interindividual variations in the endocannabinoidome mediators levels following a 2-day SFA and UFA diet intervention according to abdominal adiposity and type 2 diabetes.

SECONDARY OUTCOMES:
Gut microbiota in response to a 2 day dietary lipid intervention in abdominal obesity and type 2 diabetes | 7 days
  Interindividual variations in the gut microbiota composition following a 2-day SFA and UFA diet intervention according to abdominal adiposity and type 2 diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Veilleux, PhD, Principal Investigator — Laval University
Locations (1):
- Institut sur la nutrition et les aliments fonctionnels - INAF, Québec, Quebec, Canada